CLINICAL TRIAL: NCT04246580
Title: Evaluation of Indocyanine Green-guided Systematic Pelvic Lymphadenectomy in Endometrial and Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, Università degli Studi dell'Insubria
Other Study IDs: GREEN-1
Record Dates: First submitted 2020-01-26; First posted 2020-01-29 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Endometrial Cancer; Cervical Cancer
Keywords: Indocyanine green; Pelvic lymphadenectomy
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Indocyanine green: Women with endometrial and cervical cancer undergoing indocyanine green-guided systematic pelvic lymphadenectomy by laparoscopy or robotic surgery
  Interventions: Procedure: Indocyanine green-guided systematic pelvic lymphadenectomy
- Control: Women with endometrial and cervical cancer undergoing systematic pelvic lymphadenectomy by laparoscopy or robotic surgery without the use of indocyanine green tracer injection.

INTERVENTIONS:
Procedure: Indocyanine green-guided systematic pelvic lymphadenectomy — Injection of Indocyanine green within the uterine cervix before to perform laparoscopic/robotic systematic pelvic lymphadenectomy
  Groups: Indocyanine green

SUMMARY:
The lymph nodes involvement is one of the most important prognostic factors in endometrial (EC) and cervical cancer (CC). Indeed, the lymph node involvement in cancer patients modifies the International Federation of Gynecology and Obstetrics (FIGO) stage and plays a pivotal role in the choice of the adjuvant therapy.

Since the modern imaging techniques are not yet able to accurately detect lymph nodes metastasis, pelvic systematic lymphadenectomy has still an important role and it still represents the gold standard in EC and CC. The sentinel lymph node (SLN) biopsy, which is a standard practice in breast cancer and melanoma, is often used in some early stage gynaecological cancers such as EC and CC.

Indocyanine green (ICG) is the most used tracer for the detection of SLN in gynaecological cancer, especially in laparoendoscopic setting. ICG allows a complete visualization of the lymphatic drainage and, for this reason, it may be used even in systematic pelvic lymphadenectomy to guide the surgeon during the procedure. Several studies have demonstrated an advantage of the ICG-guided lymphadenectomy in other types of cancers, showing a higher number of lymph nodes removed with this technique when compared to standard lymphadenectomy (without ICG).

To date, there is no published study about ICG-guided systematic pelvic lymphadenectomy in EC and CC. In this scenario, the aim of this study will be to compare systematic ICG-guided pelvic lymphadenectomy and standard lymphadenectomy in EC and CC.

ELIGIBILITY:
Inclusion Criteria:

* Women affected by endometrial or cervical cancer
* Laparoscopic/robotic surgical approach with systematic pelvic lymphadenectomy.

Exclusion Criteria:

* Women undergoing open surgery (laparotomy) for the surgical management of endometrial or cervical cancer.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women affected by endometrial or cervical cancer undergoing laparoscopic/robotic systematic pelvic lymphadenectomy (with or without previous injection of indocyanine green tracer within the uterine cervix).
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Retrieved lymph nodes | At the moment of the surgery
  Number of retrieved lymph nodes after laparoscopic/robotic systematic pelvic lymphadenectomy

CONTACTS AND LOCATIONS:
Overall Officials: Benito Chiofalo, M.D., Principal Investigator — Regina Elena National Cancer Institute, Rome, Italy; Antonio Simone Laganà, M.D., Ph.D., Study Chair — Università degli Studi dell'Insubria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiofalo B, Lagana AS, Ghezzi F, Certelli C, Casarin J, Bruno V, Sperduti I, Chiantera V, Peitsidis P, Vizza E. Beyond Sentinel Lymph Node: Outcomes of Indocyanine Green-Guided Pelvic Lymphadenectomy in Endometrial and Cervical Cancer. Int J Environ Res Public Health. 2023 Feb 16;20(4):3476. doi: 10.3390/ijerph20043476. PMID 36834170